CLINICAL TRIAL: NCT01217437
Title: Temozolomide With Irinotecan Versus Temozolomide, Irinotecan Plus Bevacizumab (NSC# 704865) for Recurrent/Refractory Medulloblastoma/CNS PNET of Childhood, a COG Randomized Phase II Screening Trial
Brief Title: Temozolomide and Irinotecan Hydrochloride With or Without Bevacizumab in Treating Young Patients With Recurrent or Refractory Medulloblastoma or CNS Primitive Neuroectodermal Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02605; NCI-2011-02605 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 11-00909; CDR0000686608; COG-ACNS0821; ACNS0821; ACNS0821 (Other: Children's Oncology Group); ACNS0821 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-06

CONDITIONS: Central Nervous System Neoplasm; Pineoblastoma; Recurrent Medulloblastoma; Recurrent Primitive Neuroectodermal Tumor; Refractory Medulloblastoma; Refractory Peripheral Primitive Neuroectodermal Tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Pinealoma; Medulloblastoma; Neuroectodermal Tumors, Primitive; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Irinotecan; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (temozolomide, irinotecan hydrochloride) (Experimental): Patients receive temozolomide PO and irinotecan hydrochloride IV over 90 minutes on days 1-5.
  Interventions: Drug: Irinotecan Hydrochloride; Drug: Temozolomide
- Arm II (temozolomide, irinotecan hydrochloride, bevacizumab) (Experimental): Patients receive temozolomide PO and irinotecan hydrochloride IV as in arm I and bevacizumab IV over 30-90 minutes on days 1 and 15.
  Interventions: Biological: Bevacizumab; Drug: Irinotecan Hydrochloride; Drug: Temozolomide

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-awwb; Bevacizumab-bvzr; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; MYL-1402O; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; Zirabev
  Arms: Arm II (temozolomide, irinotecan hydrochloride, bevacizumab)
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; Irinomedac; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate; U-101440E
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This randomized phase II trial studies how well giving temozolomide and irinotecan hydrochloride together with or without bevacizumab works in treating young patients with recurrent or refractory medulloblastoma or central nervous system (CNS) primitive neuroectodermal tumors. Drugs used in chemotherapy, such as temozolomide and irinotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether temozolomide and irinotecan hydrochloride are more effective with or without bevacizumab in treating medulloblastoma or CNS primitive neuroectodermal tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

l. To compare the overall survival (OS) of subjects receiving the combination of temozolomide and irinotecan with that of subjects receiving temozolomide, irinotecan (irinotecan hydrochloride), and bevacizumab for recurrent medulloblastoma (MB)/primitive neuroectodermal tumor (PNET) of childhood.

SECONDARY OBJECTIVES:

I. To assess the response rate for each treatment arm amongst patients who are enrolled with measurable disease.

II. To determine event-free survival (EFS) for each patient compared across regimens.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive temozolomide orally (PO) and irinotecan hydrochloride IV over 90 minutes on days 1-5.

ARM II: Patients receive temozolomide PO and irinotecan hydrochloride IV as in arm I and bevacizumab IV over 30-90 minutes on days 1 and 15.

In both arms, treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Medulloblastoma or PNET of childhood that has relapsed or become refractory to standard chemotherapy; patients with pineoblastoma are eligible
* Patients must have had histologic verification of the malignancy at original diagnosis or at the time of recurrence
* Patients must have clear residual disease, defined as tumor that is measurable in two perpendicular diameters on magnetic resonance imaging (MRI) OR diffuse leptomeningeal disease OR clear MRI evidence of disease that may not be measurable in two perpendicular diameters
* All patients must have a brain MRI with and without gadolinium and a spine MRI with gadolinium performed within 2 weeks prior to study enrollment
* Patients must have a Lansky or Karnofsky performance status score of >= 50%, corresponding to Eastern Cooperative Oncology Group (ECOG) categories of 0, 1, or 2 (use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age)
* Patients must have a life expectancy of >= 8 weeks
* Patients must have experienced at least one and at most two relapses prior to study enrollment; patients with primary refractory disease are eligible
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study

  * Myelosuppressive chemotherapy: Must not have received within 3 weeks of entry onto this study (6 weeks if prior nitrosourea)
  * Biologic (anti-neoplastic agent): At least 7 days since the completion of therapy with a biologic agent; at least 3 weeks for biologic agents with a long half life, such as antibodies
  * External beam radiation therapy (XRT): Must not have received craniospinal radiotherapy within 24 weeks prior to study entry; the tumor designated as "measurable" for protocol purposes must not have received radiation within 12 weeks prior to study entry); focal radiation to areas of symptomatic metastatic disease must not be given within 14 days of study entry
  * Stem cell transplant (SCT): For autologous SCT, >= 3 months must have elapsed prior to study entry
  * Study specific limitations on prior therapy:

    * Patients must not have previously received bevacizumab, irinotecan, temozolomide or other anti-vascular endothelial growth factor (VEGF) inhibitor
    * Patients must not be taking enzyme-inducing antiepileptic medicines within 1 week of study entry
* Patients must have recovered from any surgical procedure before enrolling on this study:

  * Patients with a major surgical procedure within 28 days prior to enrollment should be excluded
  * Patients with an intermediate surgical procedure within 14 days prior to enrollment should be excluded
  * For minor surgical procedures (including Broviac line or infusaport placement), patients should not receive the first planned dose of bevacizumab until the wound is healed and at least 7 days have elapsed
  * There should be no anticipation of need for major surgical procedures during the course of the study

    * Examples of major, intermediate, or minor surgical procedures:

      * Major procedures: Major craniotomy for tumor resection; organ resection; bowel wall anastomosis; arteriovenous grafts; exploratory laparotomy; thoracotomy
      * Intermediate procedures: Ventriculoperitoneal (VP)-shunt placement; stereotactic brain biopsy
      * Minor procedures: Incision and drainage of superficial skin abscesses; punch biopsy of skin lesions; superficial skin wound suturing; bone marrow aspirate and/or biopsy; fine needle aspirations; Broviac line or infusaport placement; paracentesis or thoracocentesis
  * Please note: Lumbar punctures or placement of peripherally inserted central catheter (PICC) lines are not considered minor procedures and may occur at any time prior to or during therapy
* Hypertension must be well controlled (=< 95th percentile for age and height if patient is =< 17 years) on stable doses of medication
* Concomitant medications restrictions:

  * Growth factor(s): Must not have received within 7 days of entry onto this study
  * Steroids: Patients who are receiving corticosteroids must be on a stable or decreasing dose for at least 7 days
  * Study Specific: Patients must not be currently taking nonsteroidal anti-inflammatory drugs (NSAIDs), clopidrogel, dipyridamole or aspirin therapy > 81 mg/day
* Peripheral absolute neutrophil count (ANC) >= 1000/uL (must not have received filgrastim [G-CSF] within the prior 7 days)
* Platelet count >= 100,000/uL (transfusion independent)
* Hemoglobin >= 8.0 gm/dL (may receive packed red blood cell [PRBC] transfusions)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min OR a serum creatinine based on age/gender as follows:

  * =< 0.4 mg/dL (for patients aged 1 month to < 6 months)
  * =< 0.5 mg/dL (for patients aged 6 months to < 1 year)
  * =< 0.6 mg/dL (for patients aged 1 to < 2 years)
  * =< 0.8 mg/dL (for patients aged 2 to < 6 years)
  * =< 1 mg/dL (for patients aged 6 to < 10 years)
  * =< 1.2 mg/dL (for patients aged 10 to < 13 years)
  * =< 1.4 mg/dL (for female patients aged >= 13 years)
  * =< 1.5 mg/dL (for male patients aged 13 to < 16 years)
  * =< 1.7 mg/dL (for male patients aged >= 16 years)
* Urine protein should be screened by dipstick analysis; if protein >= 2+ on dipstick, then urine protein creatinine (UPC) ratio should be calculated; if UPC ratio > 0.5, 24-hour urine protein should be obtained and the level should be < 1000 mg/24 hours for patient enrollment
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 3 x upper limit of normal (ULN) for age
* Central nervous system function defined as

  * Patients with a seizure disorder may be enrolled if well-controlled and on non-enzyme inducing anticonvulsants
* Adequate coagulation defined as

  * International normalized ratio (INR)/prothrombin time (PT) =< 1.5 x upper limit of normal

Exclusion Criteria:

* Patients with a serious or non-healing wound, ulcer, or bone fracture are not eligible for this study
* Patients must not have a history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to study entry
* Patients must not have a known bleeding diathesis or coagulopathy
* Patients must not have had significant vascular disease (eg, aortic aneurysm requiring surgical repair, deep venous or arterial thrombosis) within the last 6 months prior to study entry
* Patients must not have a known thrombophilic condition (i.e. protein S, protein C or antithrombin III deficiency, Factor V Leiden, Factor II G20210A mutation, homocysteinemia or antiphospholipid antibody syndrome); testing is not required in patients without thrombophilic history
* Patients must not have evidence of new CNS hemorrhage on baseline MRI obtained within 14 days prior to study enrollment
* Patients with a history of stroke, myocardial infarction, transient ischemic attack (TIA), severe or unstable angina, peripheral vascular disease, or grade II or greater congestive heart failure within the past 6 months are not eligible
* Patients must not have serious and inadequately controlled cardiac arrhythmia
* Female patients who are pregnant are not eligible for this study
* Female patients who are breastfeeding are not eligible for this study unless they agree not to breastfeed
* Female patients of childbearing potential must have a negative pregnancy test
* Sexually active patients of childbearing potential must agree to use an effective method of contraception during the study and for at least 6 months after the completion of bevacizumab therapy
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Actual)
Dates: Start 2010-11-22 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam S Levy, Principal Investigator — Children's Oncology Group
Locations (158):
- United States (136):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Columbia Regional, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (7):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (12):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- University Pediatric Hospital, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Temozolomide, Irinotecan Hydrochloride) | Arm II (Temozolomide, Irinotecan Hydrochloride, Bevacizumab)
Started | 55 | 53
Completed | 12 | 12
Not Completed | 43 | 41
Not completed — Adverse Event | 0 | 8
Not completed — Death | 5 | 0
Not completed — Lack of Efficacy | 29 | 25
Not completed — Physician Decision | 8 | 5
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Ineligible | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Temozolomide, Irinotecan Hydrochloride) | Arm II (Temozolomide, Irinotecan Hydrochloride, Bevacizumab) | Total
Number analyzed (Participants) | 55 | 53 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 51 | 49 | 100
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.82 (5.29) | 10.25 (4.91) | 10.03 (5.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 37
  Male | 34 | 37 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 19
  Not Hispanic or Latino | 45 | 43 | 88
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 8 | 6 | 14
  White | 41 | 42 | 83
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 45 | 43 | 88
  Canada | 7 | 7 | 14
  Australia | 3 | 2 | 5
  New Zealand | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Percentage Probability of remaining alive 5 years after enrollment estimated by the method of Kaplan and Meier
Time Frame: Up to 5 years after enrollment
Population: Randomized eligible patients. 2 patients were excluded due to ineligibility.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Arm I (Temozolomide, Irinotecan Hydrochloride) | Arm II (Temozolomide, Irinotecan Hydrochloride, Bevacizumab)
Number analyzed (Participants) | 54 | 52
percent probability | 2.43 [0.2 to 10.9] | 13.6 [4.7 to 27.1]

2. Secondary Outcome: Response
Description: Patient's best response during protocol therapy coded as complete response, partial response or no response.
Time Frame: Up to 12 cycles of therapy (11 months)
Population: Eligible patients who were enrolled and had measurable disease according to the protocol definition at the time of enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Temozolomide, Irinotecan Hydrochloride) | Arm II (Temozolomide, Irinotecan Hydrochloride, Bevacizumab)
Number analyzed (Participants) | 48 | 46
Participants
  Complete Response | 0 | 8
  Partial Response | 16 | 14
  No Response | 32 | 24

3. Secondary Outcome: Event-free Survival
Description: Percentage Probability of remaining event-free 5 years after enrollment estimated by the method of Kaplan and Meier
Time Frame: Up to 5 years after enrollment
Population: Randomized eligible patients. 2 patients were excluded due to ineligibility.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Arm I (Temozolomide, Irinotecan Hydrochloride) | Arm II (Temozolomide, Irinotecan Hydrochloride, Bevacizumab)
Number analyzed (Participants) | 54 | 52
percent probability | 1.85 [0.15 to 8.62] | 15.4 [7.2 to 26.4]

ADVERSE EVENTS:
Time Frame: 12 cycles (planned 336 days of protocol therapy)
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution, via expedited reporting (NCI AdEERs / CAeRs). The "AE Other" table reflects all CTCAEs collected excluding those that were reported as SAEs. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Arm I (Temozolomide, Irinotecan Hydrochloride) | Arm II (Temozolomide, Irinotecan Hydrochloride, Bevacizumab)
All-Cause Mortality (participants affected / at risk) | 48/54 | 42/52
Serious Adverse Events (participants affected / at risk) | 9/54 | 12/52
Other Adverse Events (participants affected / at risk) | 31/54 | 42/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Temozolomide, Irinotecan Hydrochloride) (N=54) | Arm II (Temozolomide, Irinotecan Hydrochloride, Bevacizumab) (N=52)
Alanine aminotransferase increased (Investigations) | 1 | 1
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 1
Death NOS (General disorders) | 4 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 0 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 3 | 1
Skin infection (Infections and infestations) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
White blood cell decreased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Temozolomide, Irinotecan Hydrochloride) (N=54) | Arm II (Temozolomide, Irinotecan Hydrochloride, Bevacizumab) (N=52)
Abdominal pain (Gastrointestinal disorders) | 4 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 2
Allergic reaction (Immune system disorders) | 1 | 0
Anaphylaxis (Immune system disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 10 | 7
Anorexia (Metabolism and nutrition disorders) | 3 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 1
Ataxia (Nervous system disorders) | 1 | 0
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 2
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Creatinine increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 4
Depressed level of consciousness (Nervous system disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 13 | 15
Dysarthria (Nervous system disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Facial nerve disorder (Nervous system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 6
Fever (General disorders) | 2 | 0
GGT increased (Investigations) | 0 | 3
Headache (Nervous system disorders) | 2 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 2 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 6 | 3
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 2
Hypotension (Vascular disorders) | 4 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Infections and infestations - Other, specify (Infections and infestations) | 3 | 0
Infusion related reaction (General disorders) | 1 | 0
Lymphocyte count decreased (Investigations) | 9 | 10
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 1
Neutrophil count decreased (Investigations) | 19 | 24
Non-cardiac chest pain (General disorders) | 1 | 0
Personality change (Psychiatric disorders) | 0 | 1
Platelet count decreased (Investigations) | 15 | 19
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 2
Sepsis (Infections and infestations) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0
Sinusitis (Infections and infestations) | 0 | 2
Stomach pain (Gastrointestinal disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 1
Typhlitis (Gastrointestinal disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 7 | 2
White blood cell decreased (Investigations) | 13 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT01217437/Prot_SAP_000.pdf